CLINICAL TRIAL: NCT07121244
Title: Phase 1 Study of 68Ga-R11228 and 177Lu-R11228 in Patients With Advanced Breast Cancer
Brief Title: A Phase 1 Study of 68Ga-R11228 and 177Lu-R11228 in Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Radionetics Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R11228-101
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Locoregionally Recurrent Hormone-receptor Positive Breast Cancer; Metastatic Hormone Receptor Positive Breast Cancer
Keywords: Hormone Receptor Positive Breast Cancer; Endocrine resistant; Radioisotope

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: 68Ga-R11228 Dose Optimization Portion (Experimental): 68Ga-R11228 injection at pre-defined dose levels.
  Interventions: Drug: 68Ga-R11228
- Part B: 68Ga-R11228 Imaging and 177Lu-R11228 Dose Ranging Portion (Experimental): 68Ga-R11228 injection at pre-defined dose. 177Lu-R11228 injection at pre-defined doses.
  Interventions: Drug: 68Ga-R11228; Drug: 177Lu-R11228

INTERVENTIONS:
Drug: 68Ga-R11228 — 68Ga-R11228 is a gallium-labeled small molecule radioligand that is designed to localize tumor lesions
Drug: 177Lu-R11228 — 177Lu-R11228 is a lutetium-labeled small molecule radioligand designed to treat tumor lesions
  Arms: Part B: 68Ga-R11228 Imaging and 177Lu-R11228 Dose Ranging Portion

SUMMARY:
A phase 1 study of 68Ga-R11228 and 177Lu-R11228 in breast cancer.

DETAILED DESCRIPTION:
Patients with metastatic or locoregionally recurrent ER+ and/or PR+ and HER2 negative breast cancer will be enrolled.

Part A is being conducted to test 68Ga-R11228, a new investigational product (IP) that has been designed to detect cancer lesions in the body and make them visible on a Positron Emission Tomography (PET) scan. Three dose levels of 68Ga-R11228 will be evaluated, with each patient receiving a single dose.

Part B is being conducted to test 68Ga-R11228 and additionally 177Lu-R11228, which has been designed to treat patients who have cancer lesions with positive uptake on PET scan using 68Ga-R11228. Patients who qualify for 177Lu-R11228 treatment will receive up to 6 doses over approximately 36 weeks. Multiple 177Lu-R11228 dose levels will be evaluated in Part B.

A 5-year Follow-Up Period begins once the last cycle of 177Lu-R11228 dosing is completed.

ELIGIBILITY:
Inclusion Criteria:

Part A

* Pathologically confirmed estrogen and/or progesterone receptor (ER/PR) positive and HER2 negative locoregionally recurrent or metastatic breast cancer
* At least one target or non-target lesion per RECIST v1.1 criteria.
* Male or non-pregnant, non-lactating female subjects age ≥18 years.

Part B

* Pathologically confirmed estrogen and/or progesterone receptor (ER/PR) positive and HER2 negative locoregionally recurrent or metastatic breast cancer
* Refractory to endocrine therapy. Note: there is no limit on prior number of lines of endocrine therapy or prior treatments with CDK4/6, AKT, PI3K and/or mTOR inhibitors.
* Received or declined at least one line of chemotherapy or antibody drug conjugate in the locoregionally recurrent or metastatic setting
* Progressive disease or intolerance to last treatment.
* At least one target lesion per RECIST v1.1 criteria.
* Male or non-pregnant, non-lactating female subjects age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Life expectancy of at least six months.
* Adequate bone marrow reserve, hepatic function and renal function.

Exclusion Criteria:

Part A

* Study participant has not recovered from clinically significant adverse event(s) resulting from most recent anticancer therapy/intervention.
* Known central nervous system (CNS) disease, except for those subjects with treated brain metastasis who are stable for at least 1 month, having no evidence of progression or hemorrhage after treatment and no ongoing requirement for corticosteroids, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT]) during the screening period.
* Radiotherapy for breast cancer ≤ 28 days prior
* Received a radionuclide within a period of less than 10 physical half-lives of the administered radionuclide prior to dosing with 68Ga-R11228.
* Any condition that precludes the proper performance of imaging procedures required in this study.

Part B

* Study participant has not recovered from clinically significant adverse event(s) resulting from most recent anticancer therapy/intervention
* Treatment with anticancer therapy or with an investigational drug or device within 21 days or 5 half-lives of the agent (whichever is shorter)
* Known central nervous system (CNS) disease, except for those subjects with treated brain metastasis who are stable for at least 1 month, having no evidence of progression or hemorrhage after treatment and no ongoing requirement for corticosteroids, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT]) during the screening period.
* Radiotherapy for breast cancer ≤ 28 days
* Prior systemic radionuclide therapeutic treatment.
* Received a radionuclide within a period of less than 10 physical half-lives of the administered radionuclide prior to dosing with 68Ga-R11228.
* Any unresolved NCI-CTCAE Version 5.0 Grade 2 or higher toxicity (except alopecia and Grade 2 platinum-therapy related neuropathy) from previous breast cancer treatment and/or from medical/surgical procedures or interventions.
* Any condition that precludes the proper performance of imaging procedures required in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2033-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events [68Ga-R11228] | Day 1 to Day 7
  Number of participants with adverse events as assessed by NCI-CTCAE v5.0, including grade
Incidence of Serious Adverse Events [68Ga-R11228] | Day 1 to Day 7
  Number of participants with serious adverse events
Incidence of adverse events [177Lu-R11228] | Day 1 to week 36
  Number of participants with adverse events as assessed by NCI-CTCAE v5.0, including grade
Incidence of Serious Adverse Events [177Lu-R11228] | Day 1 to week 36
  Number of participants with serious adverse events
Incidence of dose limiting toxicities [177Lu-R11228] | Day 1 to week 36
  Number of participants with dose limiting toxicities

SECONDARY OUTCOMES:
Image quality | Day 1
  68Ga-R11228 positron emission tomography (PET) image quality as assessed by a 5-point Likert scale
Absorbed dose coefficients [68Ga-R11228] | Day 1
  Absorbed dose coefficients (milliGray [mGy]/megabecquerel [MBq]) in organs.
Standardized uptake value in tumor lesions [68Ga-R11228] | Day 1
  Standard uptake value (SUV) in tumor lesions
Effective whole-body dose for 68Ga-R11228 | Day 1
  Effective whole-body dose (millisievert [mSv]/MBq) for 68Ga-R11228
Pharmacokinetic parameters of 68Ga-R11228 | Day 1
  PK parameters, including Cmax
Pharmacokinetic parameters of 68Ga-R11228 | Day 1
  PK parameters, including area under the curve
Pharmacokinetic parameters of 68Ga-R11228 | Day 1
  PK parameters, including half-life
Pharmacokinetic parameters of 68Ga-R11228 | Day 1
  PK parameters, including total plasma clearance
Pharmacokinetic parameters of 68Ga-R11228 | Day 1
  PK parameters, including apparent volume of distribution
Pharmacokinetic parameters of 68Ga-R11228 | Day 1
  Amount of 68Ga-R11228 excreted in urine
Inter-reader agreement | Day 1
  Inter-reader agreement described by Fleiss' kappa coefficient
Intra-reader reproducibility | Day 1
  Intra-reader reproducibility described by Cohen's kappa coefficient
Number of study participants with at least one tumor lesion detected | Day 1
  Number of study participants with at least one tumor lesion detected by imaging with 68Ga-R11228
Proportion of tumor lesions detected by imaging with 68Ga-R11228 per study participant | Day 1
  Proportion of the number of tumor lesions positive with 68Ga-11228 imaging divided by the number of tumor lesions detected with standard of care images
Absorbed dose coefficients [177Lu-R11228] | 7 days
  Absorbed dose coefficients (milliGray [mGy]/megabecquerel [MBq]) in organs and tumor lesions for 177Lu-R11228
Pharmacokinetic parameters of 177Lu-R11228 | 7 days
  PK parameters, including Cmax
Pharmacokinetic parameters of 177Lu-R11228 | 7 days
  PK parameters, including area under the curve
Pharmacokinetic parameters of 177Lu-R11228 | 7 days
  PK parameters, including half-life
Pharmacokinetic parameters of 177Lu-R11228 | 7 days
  PK parameters, including total plasma clearance
Pharmacokinetic parameters of 177Lu-R11228 | 7 days
  PK parameters, including apparent volume of distribution
Objective response rate | 36 weeks
  Number of study participants with a complete or partial response divided by the number of study participants who had at least one 177Lu-11228 dose
Duration of response | 36 weeks
  Time from achieving partial response or complete response to progression per RECIST v1.1 or death, whichever is sooner
Progression free survival | 36 weeks
  Time from first 177Lu-R11228 dose until progression per RECIST v1.1 or death, whichever is sooner
Overall survival | 36 weeks
  Time from first 177Lu-R11228 dose until death from any cause

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - United Theranostics Princeton, Princeton, New Jersey
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
- Melbourne Theranostic Innovation Centre (MTIC), Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No